CLINICAL TRIAL: NCT07214649
Title: A Prospective Study Using Patient-Derived Extrahepatic Cholangiocyte Organoids for Refractory Bile Leaks
Brief Title: Organoids for Bile Leaks
Acronym: ASCORB
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, PASCALE MARCO MARIA, MD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025001; 2025001 (Registry Identifier: FPG); FPG (Other: FPG)
Record Dates: First submitted 2025-10-03; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Biliary Anastomosis Complication
Keywords: biliary leaks; cholangiocyte organoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Organoid Arm (Experimental)
  Interventions: Biological: Organoid-guided treatment

INTERVENTIONS:
Biological: Organoid-guided treatment — Engrafment of the Cholangiocyte Organoids in the common bile duct with leakage

SUMMARY:
Background: Bile leakage remains a major complication after hepatobiliary surgery and liver transplantation. While most cases are managed through standard radiologic or endoscopic interventions, a subset of patients fails to respond and may face recurrent interventions or even retransplantation. Recent advances in regenerative medicine, particularly the development of extrahepatic cholangiocyte organoids (ECOs), offer a promising alternative.

Objective: This prospective, 5-year study aims to evaluate the feasibility, safety, and efficacy of autologous ECO-based cell therapy to reconstruct bile ducts in patients with persistent bile leakage unresponsive to standard care.

Methods: Patients undergoing hepatobiliary or liver transplant surgery will have a biopsy of extrahepatic bile duct tissue collected perioperatively. The tissue will be processed and stored in a dedicated biobank. Upon development of a refractory bile leak, ECOs will be generated from the stored tissue and delivered to the site of injury through radiological or endoscopic routes, as decided by a multidisciplinary team. Success will be evaluated by resolution of leakage (radiologically or endoscopically) and absence of further intervention.

Significance: The use of patient-specific ECOs holds transformative potential. Organoids can be derived and expanded in vitro while maintaining cholangiocyte identity and function. Preclinical studies in murine and human models show successful engraftment and functional integration into biliary epithelium.

Expected Outcomes: This project aims to pioneer a novel, minimally invasive, personalized regenerative therapy for otherwise intractable biliary complications.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old
* Undergone HPB surgical procedure with hepatic duct reconstruction
* Presence of anastomotic bile leakage untreatable with radiological or endoscopic approach
* Presence of bile duct specimen

Exclusion Criteria:

* Age under 18 years old
* Undergone HPB surgical procedure without hepatic duct reconstruction
* Absence of anastomotic bile leakage untreatable with radiological or endoscopic approach
* Absence of bile duct specimen

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2030-06 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Treatment of the leaks | 1 week
  Absence of leak at radiological or endoscopic evaluation

IPD SHARING:
Plan to Share IPD: No